CLINICAL TRIAL: NCT04553835
Title: Effects of Rhythmic Auditory Stimulation on Movements in Individuals at Risk for Psychotic Onset and Schizophrenia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr WANG Shumei (Other)
Responsible Party: Sponsor-Investigator, Dr WANG Shumei, Assistant Professor, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20200630002
Record Dates: First submitted 2020-09-12; First posted 2020-09-17 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia; Psychosis; Parkinsonism; Dyskinesias
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Parkinsonian Disorders; Dyskinesias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- schizophrenia- RAS (Experimental): Schizophrenia patients in the experimental group will undergo upper-limb movement training with the aid of rhythmic auditory stimulation (RAS).
  Interventions: Behavioral: Rhythmic auditory stimulation (RAS) for schizophrenia patients
- schizophrenia- no RAS (Active Comparator): Schizophrenia patients in the control group will receive upper-limb training without the aid of RAS.
  Interventions: Behavioral: No RAS for schizophrenia patients
- at risk- RAS (Experimental): At-risk individuals in the experimental group will undergo upper-limb movement training with the aid of RAS.
  Interventions: Behavioral: RAS for at-risk individuals
- at risk- no RAS (Active Comparator): At-risk individuals in the control group will receive upper-limb training without the aid of RAS.
  Interventions: Behavioral: No RAS for at-risk individuals

INTERVENTIONS:
Behavioral: Rhythmic auditory stimulation (RAS) for schizophrenia patients — A mobile application, "metronome beats" developed by Stonekick Limited, will be used to give RAS when the participant executes the movement. Before intervention, the participant is required to execute the movement task without the aid of RAS as quickly as possible for 30 seconds, so that we obtain his/her baseline movement tempo (beats per minute). For each 40-minute training session in the first training week, three RAS tempi will be provided for the first, second, and last 10 minutes with a five-minute break in between: normal (100% of the baseline tempo), quick (105% of the baseline tempo), and fast (110% of the baseline tempo). With each training week, the three RAS tempi will be increased by 5%. Schizophrenia patients in the experimental group will undergo upper limb movement training with the aid of RAS. The intervention protocol will last for 3 weeks on the weekday basis (a total of 15 sessions) with one session (40 minutes) per weekday.
  Arms: schizophrenia- RAS
Behavioral: No RAS for schizophrenia patients — The training protocol will be the same as that used in the experimental group except the lack of RAS during execution of the movement task.
  Arms: schizophrenia- no RAS
Behavioral: RAS for at-risk individuals — A mobile application, "metronome beats" developed by Stonekick Limited, will be used to give RAS when the participant executes the movement. Before intervention, the participant is required to execute the movement task without the aid of RAS as quickly as possible for 30 seconds, so that we obtain his/her baseline movement tempo (beats per minute). For each 40-minute training session in the first training week, three RAS tempi will be provided for the first, second, and last 10 minutes with a five-minute break in between: normal (100% of the baseline tempo), quick (105% of the baseline tempo), and fast (110% of the baseline tempo). With each training week, the three RAS tempi will be increased by 5%. At-risk individuals in the experimental group will undergo upper limb movement training with the aid of RAS. The intervention protocol will last for 3 weeks on daily basis (a total of 21 sessions), with one training session (40 minutes) per day.
  Arms: at risk- RAS
Behavioral: No RAS for at-risk individuals — The training protocol will be the same as that used in the experimental group except the lack of RAS during execution of the movement task.
  Arms: at risk- no RAS

SUMMARY:
The purpose of this research is to examine effects of movement training with the aid of rhythmic auditory stimulation (RAS) on reducing severity of dyskinesia and bradykinesia in at-risk individuals and schizophrenia patients. The investigators hypothesize that training with the aid of RAS reduced severity of bradykinesia and dyskinesia in at-risk individuals as well as in schizophrenia patients.

ELIGIBILITY:
For at-risk individuals:

The inclusion criteria for at-risk individuals are:

1. A score of or above 9 in the Chinese version of the 16-item Prodromal Questionnaire (CPQ-16), or a score of or above 8.18 in the Chinese version of Community Assessment of Psychic Experiences with 15 items (CAPE-C15), or a score of or above 17 in Schizotypal Personality Questionnaire-Brief (SPQ-B);
2. A score of or above 22 in the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) to ensure that they can understand instructions;
3. A score of or above 60 in the Chinese Version of Edinburgh Handedness Inventory to ensure that they are right-handed.
4. The age ≥ 13 years.

The inclusion criteria for healthy controls are:

1. A score below the cut-off score of CPQ-16, CAPE-C15, and SPQ-B;
2. A score of or above 22 in MoCA;
3. A score of or above 60 in the Chinese Version of Edinburgh Handedness Inventory;
4. No first-degree family members having a diagnosis of mental illnesses.
5. The age ≥ 13 years.

At-risk participants and healthy controls will be excluded if they have any neurological / musculoskeletal dysfunction that may affect their upper-limb movements.

For schizophrenia patients:

The inclusion criteria for schizophrenia patients are:

1. A diagnosis of schizophrenia without other psychiatric diseases;
2. Having stable psychotic symptoms;
3. A score of or above 22 in HK-MoCA;
4. A score of or above 60 in the Chinese Version of Edinburgh Handedness Inventory.
5. The age ≥ 18 years.

The inclusion criteria for healthy controls are:

1. A score below the cut-off score of CPQ-16, CAPE-C15, and SPQ-B;
2. A score of or above 22 in MoCA;
3. A score of or above 60 in the Chinese Version of Edinburgh Handedness Inventory;
4. No first-degree family members having a diagnosis of mental illnesses.
5. The age ≥ 18 years.

Patients and healthy controls will be excluded if they have any neurological / musculoskeletal dysfunction that may affect their upper-limb movements.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right before the 1st session of the intervention
  normalized movement time (representing severity of parkinsonism). Unit: second/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right after the last session of the intervention
  normalized movement time (representing severity of parkinsonism). Unit: second/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right before the 1st session of the intervention
  normalized number of movement units (representing severity of dyskinesia). Unit: units/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right after the last session of the intervention
  normalized number of movement units (representing severity of dyskinesia). Unit: units/mm

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No